CLINICAL TRIAL: NCT04640480
Title: A Phase I, Open-Label, Dose-finding Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenously Infused SNB-101(as SN-38) in Patients With Advanced Solid Tumors
Brief Title: Dose-finding Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SNB-101(SN-38) in Patients With Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SN BioScience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNB-101-101
Record Dates: First submitted 2020-10-22; First posted 2020-11-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Breast Cancer; Pancreas Cancer; Ovarian Cancer; Small-cell Lung Cancer; Gastric Cancer; Head and Neck Cancer
Keywords: solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Small Cell Lung Carcinoma; Stomach Neoplasms; Head and Neck Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: 1-7 cohorts, dose escalation method according to modified accelerated titration design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): SNB-101 5/8mg/m2 Q2W IV
  Interventions: Drug: SNB-101
- Cohort 2 (Experimental): SNB-101 10/16mg/m2 Q2W IV
  Interventions: Drug: SNB-101
- Cohort 3 (Experimental): SNB-101 20/32mg/m2 Q2W IV
  Interventions: Drug: SNB-101
- Cohort 4 (Experimental): SNB-101 30/48mg/m2 Q2W IV
  Interventions: Drug: SNB-101
- Cohort 5 (Experimental): SNB-101 40/64mg/m2 Q2W IV
  Interventions: Drug: SNB-101
- Cohort 6 (Experimental): SNB-101 45/72mg/m2 Q2W IV
  Interventions: Drug: SNB-101
- Cohort 7 (Experimental): SNB-101 50/80mg/m2 Q2W IV
  Interventions: Drug: SNB-101

INTERVENTIONS:
Drug: SNB-101 — SN-38 dosage ranges from 1 to 7 will be determined by Safety Review Committee meeting
  Other Names: SN-38

SUMMARY:
SNB-101 is a novel nano-particle formulation of SN-38, the active metabolite of irinotecan(CPT-11). Study SNB101P01 is a multicenter, open-label, dose escalation, phase 1 study of SNB 101 with its active ingredient SN-38, in participants with advanced solid tumors. Dose escalation will occur using a modified accelerated titration design (ATD).

All participants will receive SNB 101 in different cohorts. SNB 101 will be administered intravenously to participants on day 1 and day 15 of each 28 day treatment cycle until progressive disease, unacceptable toxicity, death, or withdrawal of consent, whichever occurs first.

A Safety Review Committee will determine dose escalation, de-escalation, and modification and the MTD/RP2D based on DLTs and other safety information.

DETAILED DESCRIPTION:
Each participant will undergo a screening period, a treatment period, and a follow-up period. Participants will be followed until death, withdrawal of consent, or end of study, whichever occurs first.

During the treatment period, participants will receive SNB-101 (dose range: 5 mg/m2 to 50 mg/m2) intravenously on day 1 and day 15 of each 28 day cycle.

Dose reductions are permitted after the DLT observation period, which occurs during the first 28 days of treatment (cycle 1). Participants may permanently or temporarily (at the investigator's discretion) discontinue SNB-101. If a participant experiences a DLT or unacceptable toxicity, SNB-101 treatment should be interrupted until the observed toxicity returns to baseline or ≤ grade 1 toxicity. The start of the next cycle can be delayed up to 2 weeks at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically confirmed, locally advanced or metastatic disease, has progressed after systemic standard of care treatment for advanced disease and is not suitable for complete surgical resection.
* Patients with measurable or evaluable disease consistent with Response Evaluation Criteria in Solid Tumors version 1.1.
* Patients ambulatory with an Eastern Cooperative Oncology Group performance score of 0 or 1.
* Patients with adequate hematological, renal, and liver function(CTCAE V5.0 grade 1 or lower).
* Patients with the life expectancy of 3 months or longer.

Exclusion Criteria:

* Patients homozygous for UGT1A1*28 or UGT1A1*6 alleles.
* Patients known or suspected intolerance or hypersensitivity to main ingredient or any of the excipients of SNB-101.
* Patients with unintentional weight loss >10% within 3 months prior to screening.
* Patients who are on dialysis.
* Patients who are positive for HIVs.
* Patients with a QT interval with Fridericia's correction outside of normal.
* Patients with intestinal palsy or bowel obstruction.
* Patients with chronic inflammatory bowel disease.
* Patients who may require administration of neuromuscular blockers, peripheral muscle relaxants, etc. during the study.
* Patients who may require lapatinib during the study.
* Patients who may require attenuated vaccine during the study.
* Patients who are taking any medication that in the judgement of the investigator could have an effect on the action of SNB-101.
* Patients unable to participate in the study as judged by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | up to 18 months(depending on safety variable)
  * All participants who take at least 1 dose of SNB-101 will be assessed.
  * DLTs will be presented by dose group and the MTD determined.
    *DLTs :
    1) Hematological toxicity
  * Grade 4 thrombocytopenia
  * Grade 3 thrombocytopenia with clinically significant bleeding
  * Grade 4 neutropenia lasting > 7 days
  * ≥ grade 3 febrile neutropenia
    2) Nonhematological toxicity
  * Any ≥ grade 3 nonhematological toxicity
    3) Liver function abnormalities
  * Patients who have bone or liver metastasis with the following increases will be considered a DLT:
    1. Baseline AST or ALT = 2.5 to 5× ULN, then AST or ALT that increases to >8× ULN
    2. Baseline ALP = 2.5 to 5×ULN, then ALP increases to >8×ULN
       4) Any toxicity related to SNB-101 that results in a treatment delay of more than 2 weeks.
Permanent discontinuation of SNB-101 and dose reduction due to adverse events(AEs) | up to 18 months(depending on safety variable)
  Definition of permanent discontinuation of SNB-101:
  1. Experiencing a DLT or intolerable toxicity during the DLT observation period.
  2. Experiencing life-threatening Grade 4 adverse events (AE).
  3. Experiencing Grade 2 interstitial lung disease or Grade 4 infusion related reaction/ hypersensitivity.
     * Descriptive statistics for continuous variables, frequency and percentage for categorical variables
Number of participants with clinically meaningful changes in Laboratory test results from baseline | up to 18 months(depending on safety variable)
  * Hematology: RBC count, WBC count, hemoglobin, hematocrit, platelets, mean cell volume, mean cell hemoglobin, mean cell hemoglobin concentration, WBC differential count, ANC.
  * Serum biochemistry: BUN, creatinine, glucose (random), aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total bilirubin, total protein, albumin, Ca, P, K, Na, Cl, CO2, GGT, and LDH.
  * Coagulation: prothrombin time and international normalized ratio.
  * Viral serology: viral serology test for HIV antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus antibody. The test can be waived for participants who have results within 28 days prior to screening.
  * Urinalysis: specific gravity, protein, pH, blood, and ketones.
  * Descriptive statistics for continuous variables, frequency and percentage for categorical variables
Number of participants with clinically meaningful changes in Vital signs from baseline | up to 18 months(depending on safety variable)
  * Vital signs include blood pressure(sitSBP/sitDBP), heart rate, respiratory rate, and body temperature. Change from baseline or previous visit will be described.
  * After each infusion of SNB-101, vital signs will be monitored every 30 minutes for 3 hours on an outpatient basis.
  * Descriptive statistics for continuous variables, frequency and percentage for categorical variables
Electrocardiogram(ECG) results | up to 18 months(depending on safety variable)
  * ECG data will be collected at screening, C1D1, C3D1 and EOT.
  * ECG measurement at C1D1 and C3D1 will be performed after PK sampling at the end of the infusion (90 min.), 2.5 hours and 24 hours after drug administration.
  * ECG QT interval will be assessed for the safety endpoint(e.g. QTc prolongation)
  * Descriptive statistics for continuous variables, frequency and percentage for categorical variables
Number of clinically significant Chest radiograph findings(chest x-ray, CXR) | up to 18 months(depending on safety variable)
  * Number of clinically significant chest radiograph findings from chest x-ray.
  * Descriptive statistics for continuous variables, frequency and percentage for categorical variables

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve(AUC) | 4 months
  - The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
Maximum plasma concentration(Cmax) | 4 months
  - The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
Time to Cmax(Tmax) | 4 months
  The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
Clearance(CL) | 4 months
  The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
Volume of distribution(Vd) | 4 months
  The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
Terminal half-life(t1/2) | 4 months
  The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
Elimination rate constant | 4 months
  The PK parameter will be calculated for SN-38 based on plasma concentrations measured from the PK blood samples.
The objective response rate(ORR) | up to 18 months(depending on subject cycles)
  * Determination of the antitumor efficacy of SNB-101
  * All participants who take at least 1 dose of SNB-101 and have at least 1 post dose efficacy assessment will be assessed.
  * Computed tomography scans (abdomen/pelvic, chest) will be performed at screening and every 8 weeks (± 7 days) for tumor assessment.
  * ORR is defined as the percentage of participants who have achieved either complete response or partial response to the therapeutic intervention. Response is measured per RECIST version 1.1 as assessed by the investigator at the local site.
  * ORR will be presented as frequencies and percentages.
Disease control rate(DCR) | up to 18 months(depending on subject cycles)
  * Determination of the antitumor efficacy of SNB-101
  * All participants who take at least 1 dose of SNB-101 and have at least 1 post dose efficacy assessment will be assessed.
  * Computed tomography scans (abdomen/pelvic, chest) will be performed at screening and every 8 weeks (± 7 days) for tumor assessment.
  * DCR is defined as the percentage of participants who have achieved either complete response, partial response, or stable disease to the therapeutic intervention. Response is measured per RECIST version 1.1 as assessed by the investigator at the local site.
  * DCR will be presented as frequencies and percentages.
Overall survival(OS) | up to 18 months(depending on subject cycles)
  * Determination of the antitumor efficacy of SNB-101
  * All participants who take at least 1 dose of SNB-101 and have at least 1 post dose efficacy assessment will be assessed.
  * Computed tomography scans (abdomen/pelvic, chest) will be performed at screening and every 8 weeks (± 7 days) for tumor assessment.
  * OS is defined as the time from the first dose of SNB-101 to death from any cause.
  * OS median survival times will be calculated using the Kaplan Meier method.
Progression-free survival(PFS) | up to 18 months(depending on subject cycles)
  * Determination of the antitumor efficacy of SNB-101
  * All participants who take at least 1 dose of SNB-101 and have at least 1 post dose efficacy assessment will be assessed.
  * Computed tomography scans (abdomen/pelvic, chest) will be performed at screening and every 8 weeks (± 7 days) for tumor assessment.
  * PFS is defined as the time from the first dose of SNB-101 to documented disease progression or death due to any cause, whichever occurs earlier.
  * PFS median survival times will be calculated using the Kaplan Meier method.
Time to progression(TTP) | up to 18 months(depending on subject cycles)
  * Determination of the antitumor efficacy of SNB-101
  * All participants who take at least 1 dose of SNB-101 and have at least 1 post dose efficacy assessment will be assessed.
  * Computed tomography scans (abdomen/pelvic, chest) will be performed at screening and every 8 weeks (± 7 days) for tumor assessment.
  * TTP is defined as the time from the first dose of SNB-101 to objective tumor progression.
  * TTP will be calculated using the Kaplan Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Joohang Kim, Dr, Study Chair — CHA Medical Center at Bundang
Locations (3):
- South Korea (3):
  - CHA Medical Center, Seongnam-si, Gyeonggi-do
  - The Severance Hospital of the Yonsei University, Seoul, Seoul
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul, Seoul